CLINICAL TRIAL: NCT02972047
Title: Understanding the Pathophysiology and Effects of Diaphragmatic Breathing in Upright Gastroesophageal Reflux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Magnus Halland, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-007005
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: GERD
Keywords: Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic Breathing (Experimental): Subjects randomized to the experimental intervention arm will receive instructions and rationale for Diaphragmatic Breathing in the postprandial state and receive detailed instruction in diaphragmatic breathing.
  Following the office visit the patients with upright GERD and healthy persons will undergo a further 24 hours of pH impedance monitoring. This group will practice diaphragmatic breathing for 30 minutes after each meal.
  1. During the second 24 hour period patients with GERD and healthy persons will again consume the standard pH neutral refluxogenic meal note this with an event marker
  2. After 48 hours patients with GERD and healthy persons will present to the esophageal laboratory for probe removal
  Interventions: Behavioral: Diaphragmatic Breathing
- Life style counseling (Sham Comparator): Subjects randomized to the Sham Comparator intervention arm will engage in sham therapy (listening to music/watching TV for 30 minutes after each meal)
  Following the office visit the patients with upright GERD and healthy persons will undergo a further 24 hours of pH impedance monitoring. This group will will engage in sham therapy (listening to music/watching TV for 30 minutes after each meal)
  1. During the second 24 hour period patients with GERD and healthy persons will again consume the standard pH neutral refluxogenic meal note this with an event marker
  2. After 48 hours patients with GERD and healthy persons will present to the esophageal laboratory for probe removal
  Interventions: Behavioral: Sham Comparator

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing — Subjects in this are practice diaphragmatic breathing for 30 minutes after each meal.
  Arms: Diaphragmatic Breathing
Behavioral: Sham Comparator — Sham therapy (listening to music/watching TV for 30 minutes after each meal
  Arms: Life style counseling

SUMMARY:
This study aims to understand why patients have predominantly upright gastroesophageal reflux disease by comparing such patients to healthy persons AND whether a behavioral intervention (diaphragmatic breathing) will impact this disease

DETAILED DESCRIPTION:
There are two major patterns of gastroesophageal reflux disease (GERD), predominantly daytime and upright reflux and predominantly nocturnal and supine reflux.

Traditionally, upright reflux has been attributed to more frequent or wider opening with transient lower esophageal sphincter relaxations (TLESRs) while supine reflux results from a consistently reduced lower esophageal sphincter (LES) pressure. This may further be accounted for by the finding of larger hiatal hernias and greater pressure gradients between the crura and LES when comparing supine to upright refluxers. These findings may help explain supine reflux, but they offer little insight into the mechanisms of upright reflux.

In this study the investigators will be recruiting twenty healthy persons and up to 60 patients with GERD will be recruited from the clinical practice at Mayo Clinic Rochester. The investigators aim to study the intervention on 40 patients with GERD. However, recognizing that up to 33% of patients with typical symptoms of GERD will not have reflux by ambulatory pH monitoring (pH power of hydration), the investigators provide for enrolling up to a maximum of 60 patients which should be sufficient to yield 40 patients with upright GERD by pH monitoring. In addition, up to 10 additional healthy persons may be recruited.

Subjects with upright reflux and healthy controls will be randomized into one of two groups:

Experimental: Diaphragmatic breathing or Sham comparator: (listening to music/watching Television (TV) for 30 minutes after each meal to see how this impacts the disease.

ELIGIBILITY:
Inclusion Criteria for Healthy Persons:

-Patients 18 years of age or older with no symptoms of GERD

Inclusion Criteria for Patients:

* Patients 18 years of age or older with symptoms of GERD
* Upper gastrointestinal endoscopy within the past 6 months and a prior diagnostic pH impedance study showing predominantly upright reflux

Exclusion Criteria for Patients; Items indicated with an asterisk (*) are also exclusion criteria for healthy persons

* Patient who fulfil ROME IV Criteria for rumination disorder20
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological (e.g., spinal cord injuries, dementia, multiple sclerosis, Parkinson's disease), psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns.*
* Any prior gastric or esophageal surgery and significant intestinal or colonic resection*
* Hiatal hernia measuring 3 cm or larger as assessed by endoscopic or radiological studies
* Prior history of Los Angeles Grade C or D esophagitis, or esophageal stricture.
* Current use opioid analgesics or anticholinergic drugs.* We will permit low doses of tricyclic antidepressants, nortriptyline (up to 50 mg/day) or amitriptyline (up to 25 mg/day) provided they were commenced 3 months prior to the screening period, calcium channel or adrenergic1 antagonists
* Current use of proton pump inhibitors
* Known significant esophageal motor disorder (ie achalasia, aperistalsis, functional obstruction, jackhammer, distal esophageal spasm)*
* Inability to read due to: blindness, cognitive dysfunction, or English language illiteracy *
* Pregnant and lactating females *

Exclusion Criteria for Healthy Persons in addition to those marked with an Asterisk (*) above

* Ongoing use of Proton Pump Inhibitors ( PPIs) or a history consistent with GE reflux for 3 months or longer duration in past.
* Prior history of Los Angeles Grade B-D esophagitis
* Prior history of GERD on the basis of pH testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The total esophageal acid exposure time during the diagnostic 24hour pH study compared with the interventional study | 2 days
  The investigators will compare the total esophageal acid exposure time in minutes during the first 24 hour ambulatory pH study with the second 24 period during which patients are either randomized to biofeedback versus sham

SECONDARY OUTCOMES:
Upper gastrointestinal pressures in patients with upright GER compared to healthy people | 2 days
  Upper gastrointestinal pressures and pressure changes associated with meals will be described. Pressure differences will be measured in mmHg.
The effects of provocative maneuvers on upper gastrointestinal pressures. | 2 days
  The investigators will compare the effects of provocative maneuvers on upper gastrointestinal pressure. Pressure differences will be measured in mmHg.
The effects of provocative maneuvers on reflux | 2 days
  The investigators will compare the effects of provocative maneuvers on reflux as measured with impedance (Ohms)
The effects of diaphragmatic breathing on upper gastrointestinal pressures | 2 days
  The investigators will report any pressure changes (measures in mmHg) associated with diaphragmatic breathing on upper gastrointestinal pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Halland, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials